CLINICAL TRIAL: NCT01868659
Title: Diagnostic Time-Out: A Randomized Clinical Trial of a Checklist to Improve Diagnostic Accuracy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Iowa (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB201002794
Record Dates: First submitted 2013-05-30; First posted 2013-06-04 (Estimated); Last update posted 2016-05-11 (Estimated); Status verified 2015-05

CONDITIONS: Diagnostic Errors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Diagnostic checklist (Experimental): Diagnostic checklist used before patient discharged
  Interventions: Behavioral: Diagnostic checklist
- Usual care (Placebo Comparator): No diagnostic checklist used during patient encounter
  Interventions: Behavioral: Usual care with no diagnostic checklist

INTERVENTIONS:
Behavioral: Diagnostic checklist — Diagnostic checklist used before patient discharged
  Arms: Diagnostic checklist
Behavioral: Usual care with no diagnostic checklist — Patient receives usual care with no research intervention
  Arms: Usual care

SUMMARY:
Diagnostic errors are common, but they have been largely ignored by patient safety groups. Diagnostic errors are often traced to physicians' cognitive biases and failed heuristics (mental shortcuts). We know how these faulty thinking processes lead to diagnostic errors, but we know little about how to resist them. Faulty thinking has plagued other high-risk, high-reliability professionals, such as airline pilots and nuclear plant operators. These professions have learned from their mistakes and have developed checklists to help prevent them. The medical profession has started to use checklists and time-out periods in the operating room and intensive care unit, but these strategies have not been used to reduce diagnostic errors. The most common reason that physicians fail to make the correct diagnosis is that they never consider it. This failure could potentially be prevented if the physician took a time-out to review a checklist. Our broad long-term goal is to reduce diagnostic errors by developing interventions that help counter faulty diagnostic thinking. The specific aims of this project are to (1) determine the feasibility of taking a diagnostic time-out in the acute outpatient setting (urgent care clinic and emergency department), (2) determine if new diagnostic possibilities are seriously considered as a result of the time-out and checklist, and (3) compare the initial differential diagnosis with the new differential diagnosis following the time-out, and with the discharge diagnosis documented in the medical record, and with the "final" diagnosis based on a one-month follow-up. To achieve these aims, the investigators will ask 5 urgent-care physicians to complete a time-out procedure for 10 diagnostically challenging adult patients and 5 physicians will serve as controls (no time out) for 10 diagnostically challenging patients (total of 100 patients). The investigator will ask the intervention physicians to take a 2-minute time-out to review a complaint-specific differential-diagnosis checklist, which includes the differential diagnosis for 60 common presenting complaints, such as dyspnea and chest pain. The time-out will occur at the conclusion of the history and physical exam. We will use descriptive statistics and qualitative methods to characterize physicians' reactions to the time-out and checklists. We will use this pilot project to plan a larger study that will determine the risks and benefits of diagnostic time-outs and checklists.

DETAILED DESCRIPTION:
Diagnostic errors are common. They are more common than medication errors and they are the second leading cause of malpractice claims. They are more likely to harm patients and more likely to be preventable than other kinds of errors. Yet they have been largely ignored by patient safety groups, which have focused more on system problems than thinking problems. Diagnostic errors are often traced to physicians' cognitive biases and failed heuristics (mental shortcuts). We know how these faulty thinking processes lead to diagnostic errors, but we know little about how to resist them. Faulty thinking has plagued other high-risk, high-reliability professionals, such as airline pilots and nuclear plant operators. These professions have learned from their mistakes and have developed checklists to help prevent them. The medical profession has started to use checklists and time-out periods in the operating room and intensive care unit, but these strategies have not been used to reduce diagnostic errors. The most common reason that physicians fail to make the correct diagnosis is that they never consider it. This failure could potentially be prevented if the physician took a time-out to review a checklist. Our broad long-term goal is to reduce diagnostic errors by developing interventions that help counter faulty diagnostic thinking. The specific aims of this project are to (1) determine the feasibility of taking a diagnostic time-out in the acute outpatient setting (urgent care clinic and emergency department), (2) determine if new diagnostic possibilities are seriously considered as a result of the time-out and checklist, and (3) compare the initial differential diagnosis with the new differential diagnosis following the time-out, and with the discharge diagnosis documented in the medical record, and with the "final" diagnosis based on a one-month follow-up. To achieve these aims, the investigators will ask 5 urgent-care physicians to complete a time-out procedure for 10 diagnostically challenging adult patients and 5 physicians will serve as controls (no time out) for 10 diagnostically challenging patients (total of 100 patients). The investigator will ask the intervention physicians to take a 2-minute time-out to review a complaint-specific differential-diagnosis checklist, which includes the differential diagnosis for 60 common presenting complaints, such as dyspnea and chest pain. The time-out will occur at the conclusion of the history and physical exam. We will use descriptive statistics and qualitative methods to characterize physicians' reactions to the time-out and checklists. We will use this pilot project to plan a larger study that will determine the risks and benefits of diagnostic time-outs and checklists.

ELIGIBILITY:
Inclusion Criteria:

* Age over 18 years
* English speaking
* Being seen for acute medical problem
* Patient in family medicine or emergency room

Exclusion Criteria:

* age under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2010-04; Primary Completion 2014-11 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Diagnostic accuracy | 1 month after enrollment
  Diagnoses will be considered "correct" if the one-month followup diagnosis exactly agrees with the final diagnosis recorded in the medical record at the time of the visit. The one-month followup diagnosis will be determined by the investigators after reviewing the medical record and a one-month telephone interview with the patient. Diagnoses will be labeled "trivial discrepancy" if the one-month followup diagnosis differs in a trivial manner with the final diagnosis recorded in the medical record at the time of the visit (e.g., viral upper respiratory infection vs. viral bronchitis). Diagnoses will be labeled "important discrepancy" if the one-month followup diagnosis differs in an important manner with the final diagnosis recorded in the medical record at the time of the visit (e.g., viral bronchitis vs. bacterial pneumonia).

SECONDARY OUTCOMES:
Number of diagnoses in differential diagnosis | 1 day (At time of enrollment)
  At the conclusion of the history and physical exam, physicians will be asked for their opinion about the primary diagnosis plus any other diagnoses they believe should be considered (i.e., the differential diagnosis). The number of diagnoses in the differential diagnosis will be compared for checklist physicians vs. no-checklist physicians.

CONTACTS AND LOCATIONS:
Overall Officials: John W Ely, MD, Principal Investigator — University of Iowa